CLINICAL TRIAL: NCT05445895
Title: A Prospective, Randomized, Active-controlled, Double-blind, Parallel, Multi-center, Phase IV, Exploratory Study to Evaluate the Efficacy and Safety of Renexin CR in Patients With Acute Non-cardioembolic Ischemic Stroke
Brief Title: A Study to Evaluate the Efficacy and Safety of Renexin CR in Patients With Acute Non-cardioembolic Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNX_002
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renexin CR 200/160mg (Experimental): Renexin CR 200/160mg will be added to Aspirin 100mg
  Interventions: Drug: Renexin CR 200/160mg
- Clopidogrel 75mg (Active Comparator): Plavix 75mg will be added to Aspirin 100mg
  Interventions: Drug: Plavix 75mg

INTERVENTIONS:
Drug: Renexin CR 200/160mg — Renexin CR 200/160mg will be added to Aspirin 100mg
  Arms: Renexin CR 200/160mg
Drug: Plavix 75mg — Plavix 75mg will be added to Aspirin 100mg
  Arms: Clopidogrel 75mg

SUMMARY:
A study to Evaluate the Efficacy and Safety of Renexin CR in patients with Acute Non-cardioembolic Ischemic Stroke

ELIGIBILITY:
Inclusion Criteria:

1) Patients identified as acute non-cardioembolic ischemic stroke on MRI within 72 hours of onset of symptoms of cerebral infarction.

Exclusion Criteria:

1. Patients with active cancer; vascular malformation, abscess, or other major non-ischemic brain disease (e.g., multiple sclerosis).
2. With a modified Rankin Score (mRS) of 3 or higher before onset.
3. Underwent intravenous thrombolytic therapy (intravenous rtPA) or mechanical thrombectomy within 24 hours of the screening visit.
4. History of hypersensitivity to IP or components
5. Not suitable for aspirin administration at the discretion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
- The sum of the rate of neurological deterioration during hospitalization after taking the IP and the rate of stroke up to 90 days | up to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ha SH, Lee YB, Kang HG, Choi KH, Kim BJ, Woo HG, Kwon HS, Song TJ, Kim BJ. Rationale and design of the efficacy and safety of combination of cilostazol and gingko biloba extract EGb 761 in patients with acute non-cardioembolic ischemic stroke (RENEW): A pilot and feasibility randomized controlled trial. J Stroke Cerebrovasc Dis. 2025 Jan;34(1):108105. doi: 10.1016/j.jstrokecerebrovasdis.2024.108105. Epub 2024 Nov 10. PMID 39528058